CLINICAL TRIAL: NCT04580290
Title: The JewelACL Post Market Clinical Follow Up Study - Multicentre Study of at Least 5 Years Follow up, Looking at Clinical Outcomes in Patients Treated With the JewelACL for Anterior Cruciate Ligament (ACL) Reconstruction
Brief Title: Jewel ACL Post Market Clinical Follow Up Study
Status: Completed | Type: Observational
Sponsor: Xiros Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CRE 027
Record Dates: First submitted 2020-10-05; First posted 2020-10-08 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- JewelACL + Autograft (Hybrid): JewelACL + Autograft (Hybrid)
  Interventions: Device: JewelACL
- JewelACL only: JewelACL only
  Interventions: Device: JewelACL

INTERVENTIONS:
Device: JewelACL — The JewelACL is a polyester scaffold for anterior cruciate ligament (ACL) reconstruction

SUMMARY:
The objective of the study is to assess re-rupture rates and patient outcomes from subjects with at least 5 year follow up, treated with the JewelACL device for ACL reconstruction. The impact of fixation type and autograft augmentation will also be assessed. All adverse events related to the JewelACL device will be recorded. This study is Sponsored by Xiros.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Patients previously implanted with the JewelACL for Anterior Cruciate Ligament (ACL) reconstruction (Primary JewelACL cases only, no revision cases)

Exclusion Criteria:

* Age less than 18 years
* Any implantations for non-indicated conditions, as stated in the Instructions For Use Instructions for use (IFU)
* Revision cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who have had the JewelACL device used to reconstruct the ACL, between the period of 01 October 2010 to 31 December 2014.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Med-Polonia, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- JewelACL Only: Patients who received JewelACL only
- JewelACL + Autograft (Hybrid): Patients who received a JewelACL and autograft
Period: Overall Study
Arm/Group | JewelACL Only | JewelACL + Autograft (Hybrid)
Started | 88 | 32
Completed | 88 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Jewel ACL Only: Subjects who received only the JewelACL
- JewelACL + Autograft (Hybrid): Subjects who received the JewelACL + Autograft (hybrid)
- Total: Total of all reporting groups
Arm/Group | Jewel ACL Only | JewelACL + Autograft (Hybrid) | Total
Number analyzed (Participants) | 88 | 32 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (10.1) | 32.2 (11.4) | 32.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 5 | 22
  Male | 71 | 27 | 98
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Sports participation-yes [Count of Participants; unit: Participants] | 66 | 24 | 90
Cause of ACL failure [Count of Participants; unit: Participants]
  Sports Injury | 72 | 23 | 95
  Traffic Accident | 3 | 1 | 4
  Other Accident | 3 | 4 | 7
  Not available | 10 | 4 | 14
Femoral Fixation [Count of Participants; unit: Participants]
  Endobutton TightRope Arthrex | 0 | 1 | 1
  Linvatec XO | 0 | 1 | 1
  Medgal Screw | 86 | 29 | 115
  S+N EndoButton | 2 | 1 | 3
Tibial Fixation Medgal screw [Count of Participants; unit: Participants] | 88 | 32 | 120

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Re-ruptures
Description: Number of participants with re-rupture that were implanted with the jewelACL device for ACL reconstruction
Time Frame: Five Year
Measure: Count of Participants; unit: Participants
Arm/Group | JewelACL Only | JewelACL + Autograft (Hybrid)
Number analyzed (Participants) | 88 | 32
Participants | 5 | 1

ADVERSE EVENTS:
Time Frame: From time of surgery to the minimum follow up period (5 years post surgery)
Description: AE: Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs, in subjects, users or other persons, in the context of a clinical investigation, whether or not related to the investigational device.
  SAE: Any AE that led to: death,serious deterioration in the health of the subject, permanent impairment to a body structure or a body function,chronic disease,foetal distress, foetal death or a congenital physical or mental impairment or birth defect
Arm/Group | JewelACL Only | JewelACL + Autograft (Hybrid)
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/32
Serious Adverse Events (participants affected / at risk) | 5/88 | 1/32
Other Adverse Events (participants affected / at risk) | 1/88 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JewelACL Only (N=88) | JewelACL + Autograft (Hybrid) (N=32)
Rupture (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) — Re-Rupture of the ACL
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JewelACL Only (N=88) | JewelACL + Autograft (Hybrid) (N=32)
Infection (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Decreased ROM identified. Later knee pain, tests results showed infection

LIMITATIONS AND CAVEATS:
Reruptures can be sustained during sports trauma and cannot necessarily be attributed to device insufficiency.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT04580290/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT04580290/SAP_001.pdf